CLINICAL TRIAL: NCT04694508
Title: Intraoperative Music Therapy for the Reduction of Postoperative Pain in Patients Undergoing an Enhanced Recovery After Surgery Protocol in Gynecological Oncology : A Randomized Controlled Trial.
Brief Title: Intraoperative Music Therapy in Gynecological Oncology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ID-RTF065
Record Dates: First submitted 2020-12-11; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Music Therapy; General Anesthesia; Surgery; Pain; Gynecological Cancer; Pain, Postoperative
MeSH Terms: conditions — Pain; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned to either receiving intraoperative music therapy (Group A) or undergoing standard management without music therapy (Group B). Randomization was performed by a nurse specialist blinded to the study using anonymized, opaque envelopes provided by the Vall d'Hebron Research Institute. Participants were then randomized (i.e. given an envelope) to either Group A or Group B during the preoperative visit. The randomization allocation was performed using the ralloc function in STATA which randomly assigned participants in either of the two study groups in blocks of 2, 4, 6, until the total number of patients was achieved (n = 80).
Masking Description: Music therapy was administered before initiating anesthetic induction with the patient lying flat on the surgical table. A pair of non-reusable headphones (Disok, Alicante, Spain) were used in both groups which were connected to a tablet Fire 7 (Amazon, Seattle, WA, US) that was used as a music player device connected to Spotify. Two music lists were downloaded and reproduced without the need of access to WIFI to ensure good reproducibility. Group A was played a list consisting of rhythmic tones of 60-80bpm, music from the Seatwork 60bpm playlist with a duration of 11h and 5 minutes. Group B was played an empty playlist. Volume was set at a standard of 68dB. The surgical supervisor was responsible for opening the opaque envelope for each patient and to play the list according to the allocated group. Only the surgical supervisor knew the allocation for each patient, the rest of the surgical team were blinded to the allocation result.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Headphones (Disok, Alicante, España)
  Interventions: Device: Headphones (Disok, Alicante, España)
- Group B (No Intervention): Without music therapy

INTERVENTIONS:
Device: Headphones (Disok, Alicante, España) — A pair of non-reusable headphones (Disok, Alicante, Spain)
  Arms: Group A

SUMMARY:
Background Perioperative anxiety and postoperative pain can impact surgical morbidity. We aimed to evaluate the effect of intraoperative music therapy in the reduction of immediate postoperative pain in patients undergoing gynecological oncology surgery within an Enhanced Recovery After Surgery (ERAS) protocol. Secondary objectives include reduction in preoperative anxiety, postoperative pain overtime, neurohormonal response, morbidity, length of hospital stay (LOS) and patient satisfaction.

Methods Prospective, randomized, double-blinded single-center study including patients undergoing surgery for ovarian, endometrial or cervical cancer over a period of 12 months. Patients were randomly assigned to receiving intraoperative music therapy (Group A) or undergoing standard management (Group B). A reduction in immediate postoperative pain was defined as a reduction in ≥2 points in the Verbal Rating Scale(VRS) at 4h postoperatively. Hemodynamic variables and blood samples were collected during the procedure for determination of cortisol levels. A scale of closed numeric questions (Likert-like) was used to assess patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing gynecological oncology surgery for ovarian, endometrial or cervical cancer by laparotomy, laparoscopy or robotic surgery.
* ASA grade I-III
* Signed an informed consent prior to inclusion

Exclusion Criteria:

* ASA IV
* Active ischemic cardiopathy
* Hearing impairment
* Hormonal disfunction
* Active treatment with steroids
* Ppsychiatric disorder
* Contraindication for epidural anesthesia or failure of the technique in the peri-operative period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This is a clinical trial that enrolled all patients undergoing gynecological oncology surgery for ovarian, endometrial or cervical cancer by laparotomy, laparoscopy or robotic surgery.
Enrollment: 80 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

PRIMARY OUTCOMES:
The reduction in postoperative pain in patients undergoing gynecological oncology surgery within the ERAS protocol with the use of music therapy. | 1 year
  The main objective of this study was to evaluate the reduction in postoperative pain, defined as a reduction in two or more points in the VRS, in patients undergoing gynecological oncology surgery within the ERAS protocol with the use of music therapy. VRS is verbal rating score is a numeric rating scale (NRS-11) is an 11-point scale for patient self-reporting of pain. 0 means you have no pain; one to three means mild pain; four to seven is considered moderate pain; eight and above is severe pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Sánchez-Migallón Pérez, Barcelona, Spain